CLINICAL TRIAL: NCT02170467
Title: Study of Intestinal Permeability in Patients With Anorexia Nervosa
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012/174/HP
Record Dates: First submitted 2014-04-03; First posted 2014-06-23 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Anorexia Nervosa
Keywords: Intestinal permeability - Anorexia nervosa- Re feeding - auto-antibodies α-MSH
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental): Assessment of intestinal permeability in small intestine (Lactulose/ Mannitol ratio) in controls and camparison with pateints with anorexia nervosa.
  Interventions: Other: assessment of the intestinal permeability
- patients with anorexia nervosa (Experimental): Assessment of intestinal permeability in small intestine (Lactulose/ Mannitol ratio) in patients with anorexia nervosa before and after re-feeding.
  Interventions: Other: assessment of the intestinal permeability

INTERVENTIONS:
Other: assessment of the intestinal permeability

SUMMARY:
In healthy humans, the intestinal mucosa acts as an absorption organ and a defensive barrier preventing the passage of toxic substances from the intestinal lumen to the blood stream. Malnutrition and absence of exogenous luminal nutrients in the gastrointestinal tract profoundly affect small bowel morphology and physiology. Many reports have described alterations of ion and nutrient transport, mucosal atrophy and modifications in the intestinal permeability to macromolecules in cases of prolonged intestinal rest, as in severe starvation. These changes may dampen both the absorptive and the barrier functions of intestinal mucosa.

The assessment of intestinal permeability, by measuring the urinary excretion of substances that are not metabolised by human tissues and passively cross the intestinal epithelium, is a reliable and non invasive method to investigate the anatomo-functional integrity of the intestinal mucosa. Previous studies have shown an increase of permeability in malnourished humans . The increase of may also increase the risk for inappropriate passage of food antigens and other noxious substances across the mucosal barrier. To this regard, the enhanced susceptibility of malnourished subjects to systemic infections and postoperative sepsis has long been recognised.

Anorexia nervosa is a psychiatric disorder characterised by abnormal eating behaviours aiming to decrease body weight. Typically, women with anorexia nervosa restrict food ingestion up to severe starvation. These behaviours usually lead to malnutrition and a more or less prolonged absence of luminal nutrients in the gastrointestinal tract. Therefore, alterations in the integrity and functioning of intestinal mucosa are likely to occur in this condition. There is no information on intestinal permeability in patients with eating disorders. We hypothesised that, as it occurs in simple starvation and malnutrition, intestinal permeability should be increased in fasted undernourished people with anorexia nervosa and decrease after re feeding. Therefore, in the present study, we explored intestinal permeability of 23 subjects with anorexia nervosa by means of the lactulose-mannitol test and urinary sucralose excretion and compare them to 46 controls.

Moreover, auto-antibodies (α-MSH ) have been found in patients with anorexia nervosa. The origin of these auto-antibodies is still unknown , but some studies suggested a digestive origin. Moreover, modifications of intestinal flora have been described in patients with anorexia nervosa. Actually, a study of the intestinal barrier of patients with anorexia nervosa is necessary. In this study, a comparaison of intestinal permeability and autoantibodies (α-MSH) rate is proposed before and after re-feeding in patients with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

Patients with anorexia nervosa :

* female,
* living in Upper Normandy since 1 year at least,
* between 18 and 50 years of age
* with a BMI between 14 and 16 kg/m²,
* diagnosed as anorexia nervosa according to the DSM IV criteria
* hospitalised for the first time in the Nutrition Unit
* not being pregnant (effective contraception and negative pregnancy test)
* not breast-feeding,
* HIV-1 negative ,
* HIV-2 negative,
* HBV negative (hépatitis B virus),
* HCV negative (hépatitis C virus),
* Affiliated to the National Health Service,
* Giving a filled informed consent,
* Not included in other studies

Controls :

* female,
* living in Upper Normandy since 1 year at least,
* between 18 and 50 years of age,
* with a BMI between 20 and 24,9 kg/m²,
* without antecedent or current diagnosis of eating disorders (DSM IV criteria),
* without dyspepsia or irritable bowel syndrom for 6 month,
* not being pregnant (effective contraception and negative pregnancy test)
* not breast-feeding,
* HIV-1 negative ,
* HIV-2 negative,
* HBV negative (hépatitis B virus),
* HCV negative (hépatitis C virus),
* Affiliated to the National Health Service,
* Giving a filled informed consent,
* Not included in other studies

Exclusion Criteria:

Patients with anorexia nervosa :

* Adult under guardianship,
* Patient with inflammatory bowel disease and/or psychotic disorders,
* Antecedent of digestive surgery,
* Drug addiction for the last 6 month,
* Alcohol and/or other substance use disorder,
* Current immunological treatment, and/or non steroidal anti inflamatory and/or corticosteroids and/or anticoagulants and/or platelet antiaggregants
* galactosemia
* Lactulose intolerance,
* Laxatives intake in the last 3 days
* Antecedent of digestive surgery,

Controls :

* Adult under guardianship,
* Patient with inflammatory bowel disease and/or psychotic disorders,
* Antecedent of digestive surgery,
* Drug addiction for the last 6 month,
* Alcohol and/or other substance use disorder,
* Current immunological treatment, and/or non steroidal anti inflamatory and/or corticosteroids and/or anticoagulants and/or platelet antiaggregants
* galactosemia
* Lactulose intolerance,
* Laxatives intake in the last 3 days
* Antecedent of digestive surgery,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-01-05; Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
% of Sugar urinary excretion | From day 1 to Day 17, assessment after a 10% weight gain under renutrition
  intestinal permeability test - oral intake of lactulose - mannitol - sucralose

SECONDARY OUTCOMES:
sucralose urinary sampling | From day 1 to Day 17, assessment after a 10% weight gain under renutrition
  colon permeability assessement

OTHER OUTCOMES:
Evolution of auto-antibodies level ((a-MSH) after re-feeding in patients with anorexia nervosa | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien GRIGIONI, MD, Study Chair — CHU-Hôpitaux de Rouen
Locations (2):
- France (2):
  - Hôpital de la Croix Rouge, Bois-Guillaume
  - CHU- Hôpitaux de Rouen, Rouen